CLINICAL TRIAL: NCT00505570
Title: Percutaneous Closure of Patent Foramen Ovale In Migraine With Aura - A Randomized Prospective Study (Prima Trial)
Brief Title: PRIMA PFO Migraine Trial
Acronym: PRIMA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AGA010E
Record Dates: First submitted 2007-07-20; First posted 2007-07-23 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Migraine; Migraine With Aura; Patent Foramen Ovale; PFO
Keywords: Migraine; Migraine with aura; Patent foramen ovale; PFO
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Foramen Ovale, Patent

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Management (No Intervention)
- PFO Closure (Experimental)
  Interventions: Device: AMPLATZER® PFO Occluder Device

INTERVENTIONS:
Device: AMPLATZER® PFO Occluder Device — PFO device closure
  Arms: PFO Closure

SUMMARY:
The purpose of this study is to evaluate migraine headache frequency in subjects who have migraine with aura and a patent foramen ovale (PFO, a slit-like opening between the right and left upper chambers (atria) of the heart which normally closes at or soon after birth) who are randomized to either undergo closure of the patent foramen ovale or continue with standard medical management.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate migraine headache frequency in subjects who have migraine with aura and a patent foramen ovale (PFO, a slit-like opening between the right and left upper chambers (atria) of the heart which normally closes at or soon after birth) who are randomized to either undergo closure of the patent foramen ovale or continue with standard medical management.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are age 18 to 65
* Subjects who have migraine headaches with aura diagnosed by a doctor
* Subjects who have not responded to or cannot take common migraine preventive medications

Exclusion Criteria:

* Subjects with a clinical history of stroke
* Subjects who cannot take aspirin and clopidogrel (Plavix)
* Subjects who are pregnant or desire to become pregnant within the next year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Migraine headache frequency | 12 months

SECONDARY OUTCOMES:
Responder rate; Acute migraine medication use; Quality of life evaluations; Effects of Anti-thrombotic medications; Adverse events; PFO Closure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Prima Trial Steering Committee, Study Chair
Locations (17):
- Canada (7):
  - University of Calgary- Foothills Hospital, Calgary, Alberta
  - Alberta Health Services and the University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - University of Ottawa, Ottawa, Ontario
  - Davisville Medical Center, Toronto, Ontario
  - Institut de Cardiologie de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Québec, Québec, Quebec
- Germany (5):
  - Unfallkrankenhaus Berlin, Berlin
  - Martin-Luther-University Halle-Wittenberg, Halle
  - Universitätsklinikum Hamburg, Hamburg
  - Neurologisch-verhaltensmedizinische Schmerzklinik Kiel, Kiel
  - Universitätsklinikum Münster, Münster
- Switzerland (2):
  - Swiss Cardiovascular Center Bern, Bern
  - Kopfwehzentrum Hirslanden Zürich, Zurich
- United Kingdom (3):
  - Royal Sussex County Hospital, Brighton
  - St. Mary's Hospital Imperial College Healthcare NHS Trust, London
  - South Manchester University Hospital, Manchester

REFERENCES:
- [Derived] Mattle HP, Evers S, Hildick-Smith D, Becker WJ, Baumgartner H, Chataway J, Gawel M, Gobel H, Heinze A, Horlick E, Malik I, Ray S, Zermansky A, Findling O, Windecker S, Meier B. Percutaneous closure of patent foramen ovale in migraine with aura, a randomized controlled trial. Eur Heart J. 2016 Jul 7;37(26):2029-36. doi: 10.1093/eurheartj/ehw027. Epub 2016 Feb 22. PMID 26908949